CLINICAL TRIAL: NCT04428476
Title: Open-Label Extension of the HOPE-2 Duchenne Muscular Dystrophy Trial
Brief Title: Open-label Extension of the HOPE-2 Trial
Acronym: HOPE-2-OLE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Capricor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAP-1002-DMD-02-OLE
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD, Muscular dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: Open Label Extension of the HOPE-2 Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Deramiocel (Other): Participants will receive an intravenous (IV) infusion of deramiocel (150 million Cardiosphere-Derived Cells (CDCs) per infusion) every 3 months
  Interventions: Biological: Deramiocel (CAP-1002)

INTERVENTIONS:
Biological: Deramiocel (CAP-1002) — Peripheral infusion of 150 million allogeneic cardiosphere-derived cells administered every three months
  Other Names: Allogeneic Cardiosphere-Derived Cells

SUMMARY:
This Phase 2, multi-center, open-label extension trial will provide deramiocel (CAP-1002) to subjects that were enrolled in the HOPE-2 trial and completed 12 months of follow-up. The trial will explore the safety and efficacy of twenty intravenous administrations of deramiocel, each separated by three months, over a period of approximately 60 months. Following completion of the initial open-label phase (Month 60), subjects who have completed all Month 60 assessments will be eligible to continue into a long-term open label extension (LT-OLE) period and can continue to receive deramiocel once every 3 months until deramiocel is commercially available or the sponsor terminates the study, or the subject withdraws consent or study participation is terminated by the sponsor.

Subjects will undergo a targeted screening during a 30-day screening period, eligible subjects will then undergo baseline safety and efficacy assessments on Day 1 prior to their first infusion of deramiocel.

Subjects will complete trial assessments at Screening; Day 1; Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, and all LT-OLE visits. Safety and efficacy assessments will be conducted prior to deramiocel administration at the Day 1, Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, and at all LT-OLE trial visits, unless otherwise indicated.

All deramiocel infusions will be conducted in an outpatient setting at the investigative site on Day 1 and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, with continued dosing in the LT-OLE visits. Subjects will be observed in the outpatient setting for at least two hours post infusion and then discharged the same day, if medically cleared by the site Investigator.

DETAILED DESCRIPTION:
This Phase 2, multi-center, open-label extension trial will provide deramiocel (CAP-1002) to subjects that were enrolled in the HOPE-2 trial and completed 12 months of follow-up. The trial will explore the safety and efficacy of twenty intravenous administrations of deramiocel, each separated by three months, over approximately a period of 60 months. Additional analyses of efficacy and safety will be conducted in the subsequent Long Term Open-Label Extension (LT-OLE) phase of the study.

Subjects will undergo a targeted screening during a 30-day screening period to determine eligibility based on protocol inclusion and exclusion criteria.

Eligible subjects will undergo baseline safety and efficacy assessments on Day 1 prior to their first infusion of deramiocel. Administration of deramiocel (Day 1) should occur within a maximum of 30 days following confirmation of eligibility.

Subjects will complete trial assessments at Screening; Day 1; Months 3, 6, 9, 12 (± 14 days, each), 15, 18, 21, 24, 27, 30, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, and all LT-OLE visits (± 21 days, each). Safety and efficacy assessments will be conducted prior to deramiocel administration at the Day 1, Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, and 57 trial visits, unless otherwise indicated, and at all LT-OLE visits.

All deramiocel infusions will be conducted in an outpatient setting at the investigative site on Day 1 and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57 trial visits. Continued dosing in the LT-OLE phase will begin at LT-OLE Visit 1, which may overlap with Month 60 of the initial OLE phase/LT-OLE Visit 1, in some cases. Prior to each deramiocel administration, medications will be administered to the subject as determined by the Investigator based on the pre-treatment guidelines as outlined in the protocol and/or institutional protocols to minimize the risk of potential severe allergic reactions such as anaphylaxis. Subjects will be observed in the outpatient setting for at least two hours post infusion and then discharged the same day if medically cleared by the site Investigator. If clinically indicated, an unscheduled in-person visit will be performed at the investigative site with targeted assessments based on presentation of signs and symptoms following any infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Documented enrollment in the HOPE-2 trial and completion of trial follow-up through Month 12
2. Willing and able to provide informed consent to participate in the trial if ≥ 18 years of age, and assent with parental or guardian informed consent if < 18 years of age
3. Adequate venous access for intravenous deramiocel (CAP-1002) infusions in the judgement of the Investigator
4. Assessed by the Investigator as willing and able to comply with the requirements of the trial

Exclusion Criteria:

1. Planned or likely major surgery in the next 12 months after planned first infusion
2. Risk of near-term respiratory decompensation in the judgment of the investigator, or the need for initiation of non-invasive ventilator support as defined by serum bicarbonate ≥ 29 mmol/L
3. History of non DMD-related chronic respiratory disease including, but not limited to, asthma, bronchitis, and tuberculosis
4. Acute respiratory illness within 60 days prior to first infusion
5. Known hypersensitivity to dimethyl sulfoxide (DMSO) or bovine products
6. Treatment with an investigational product ≤ 6 months prior to first infusion
7. History, or current use, of drugs or alcohol that could impair ability to comply with participation in the trial
8. Inability to comply with the investigational plan and follow-up visit schedule for any reason, in the judgment of the investigator

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2026-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Craig McDonald, MD, Principal Investigator — UC Davis; Mark Awadalla, Study Director — Capricor Inc.
Locations (5):
- United States (5):
  - University of California, Davis, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Deramiocel: Participants will receive an intravenous (IV) infusion of deramiocel (150 million Cardiosphere-Derived Cells (CDCs) per infusion) every 3 months for total of 20 IV infusions.
Period: Overall Study
Arm/Group | Deramiocel
Started | 13
Completed | 0
Not Completed | 13
Not completed — Withdrawal by Subject | 1
Not completed — Still on treatment | 12

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received investigational product.
Groups:
- Deramiocel: Participants will receive an intravenous (IV) infusion of deramiocel (150 million Cardiosphere-Derived Cells (CDCs) per infusion) every 3 months for a total of 20 IV infusions.
Arm/Group | Deramiocel
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) From Baseline Through Month 12
Description: Adverse event (AE) is defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after the treatment start date. TEAEs included both serious and non-serious TEAEs.
Time Frame: Baseline up to Month 12
Population: Safety population included all participants who received investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Deramiocel
Number analyzed (Participants) | 13
Participants | 11

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity From Baseline Through Month 12
Description: Severity of adverse events (AE) were assessed by the investigator as Grade 1 = Mild (Transient or mild discomfort; no limitation in activity; no medical intervention/therapy required), Grade 2 = Moderate (Mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required), Grade 3 = Severe (Marked limitation in activity, some assistance usually required; medical intervention/therapy required and often requiring hospitalization or prolongation of hospitalization), Grade 4 = Life-threatening (Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required; hospitalization, prolongation of hospitalization, or hospice care) and Grade 5 = Death.
Time Frame: Baseline up to Month 12
Population: Safety population included all participants who received investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Deramiocel
Number analyzed (Participants) | 13
Participants
  Grade 1 | 6
  Grade 2 | 3
  Grade 3 | 2
  Grade 4 | 0
  Grade 5 | 0

3. Primary Outcome: Change From Baseline in Functional Capacity as Assessed by Performance of the Upper Limb Test, Version 2 (PUL 2.0) Total Score.
Description: PUL 2.0 scale is a 22-item scale used to assess the change that occurs in motor performance of the upper limb overtime from when a participant is still ambulant to the time participant loses all arm function when non-ambulant. PUL 2.0 includes an entry item to define broad starting functional level and 22 items subdivided into shoulder level (six items), mid-level (nine items), and distal level (seven items). Each dimension (shoulder, mid, distal) can be scored separately. There is maximum score of 12 for shoulder level, 17 for mid-level, and 13 for distal level. The total score was calculated by adding three level scores and ranged from 0-42. Higher score indicates better upper limb function.
Time Frame: Baseline, Month 12
Population: Safety population included all participants who received investigational product.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deramiocel
Number analyzed (Participants) | 13
units on a scale | -1.8 (3.07)

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) at Month 24, Month 36, Month 48 and Month 60
Description: as for outcome 1
Time Frame: Month 24, Month 36, Month 48 and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity From Baseline Through Month 60
Description: as for outcome 2
Time Frame: Baseline up to Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

6. Secondary Outcome: Change From Baseline in Upper Limb Function as Assessed by Performance of the Upper Limb Test, Version 2 (PUL 2.0) at Month 12, Month 24, Month 36, Month 48, and Month 60
Description: as for outcome 3
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

7. Secondary Outcome: Change From Baseline in Distal-Level (Wrist and Hand) Upper Limb Function as Assessed by Performance of the Upper Limb Test, Version 2 (PUL 2.0) at Month 12, Month 24, Month 36, Month 48, and Month 60
Description: as for outcome 3
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

8. Secondary Outcome: Change From Baseline in Mid-Level (Elbow) as Assessed by Performance of the Upper Limb Test, Version 2 (PUL 2.0) at Month 12, Month 24, Month 36, Month 48, and Month 60
Description: as for outcome 3
Time Frame: Baseline, Month 12, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

9. Secondary Outcome: Change From Baseline in Cardiac Parameter: Left Ventricular Ejection Fraction (LVEF) at Month, 24, 36, 48, and 60
Description: LVEF is a measurement of how much blood the left ventricle pumps out with each contraction. Change in LVEF from baseline as measured by Cardiac Magnetic Resonance (cMRI)
Time Frame: Baseline, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

10. Secondary Outcome: Change From Baseline in Cardiac Parameter: Left Ventricular End Systolic Volumes-Indexed (LV-ESVI) at Month 24, Month 36, Month 48, and Month 60
Description: Change from baseline in LV-ESVI as assessed by Cardiac Magnetic Resonance (cMRI).
Time Frame: Baseline, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

11. Secondary Outcome: Change From Baseline in Cardiac Parameter: Left Ventricular End Diastolic Volumes-Indexed (LV-EDVI) at Month 24, Month 36, Month 48, and Month 60
Description: Change from baseline in LV-EDVI as assessed by Cardiac Magnetic Resonance (cMRI.
Time Frame: Baseline, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

12. Secondary Outcome: Change From Baseline in Cardiac Parameter: Left Ventricle Mass (LV Mass) at Month 24, Month 36, Month 48, and Month 60
Description: Change from baseline in LV mass was assessed by Cardiac Magnetic Resonance (cMRI).
Time Frame: Baseline, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

13. Secondary Outcome: Change From Baseline in Cardiac Parameter: Unindexed Volumes at Month 24, Month 36, Month 48, and Month 60
Description: Change from baseline in unindexed volumes as assessed by Cardiac Magnetic Resonance (cMRI)
Time Frame: Baseline, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

14. Secondary Outcome: Change From Baseline in Cardiac Parameter: Left Ventricle End Diastolic Wall Thickening (LVEDWT) at Month 24, Month 36, Month 48, and Month 60
Description: Change from baseline in LVEDWT was assessed by Cardiac Magnetic Resonance (cMRI).
Time Frame: Baseline, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

15. Secondary Outcome: Change From Baseline in Cardiac Parameter: Left Ventricle End Systolic Wall Thickening (LVESWT) at Month 24, Month 36, Month 48, and Month 60
Description: Change from baseline in LVESWT was assessed by Cardiac Magnetic Resonance (cMRI).
Time Frame: Baseline, Month 24, Month 36, Month 48, and Month 60
Reporting Status: Not Posted, anticipated posting 2027-05

ADVERSE EVENTS:
Time Frame: Up to Month 12
Arm/Group | Deramiocel
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 11/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deramiocel (N=13)
Cardiac Dysfunction (Cardiac disorders) | 2
Supraventricular Extrasystoles (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular Extrasystoles (Cardiac disorders) | 1
Secondary Hypogonadism (Endocrine disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 3
Eyelid Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis Streptococcal (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Ligament Injury (Injury, poisoning and procedural complications) | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Heart Rate Increased (Investigations) | 1
Respiratory Rate Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Deformity Thorax (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2
Mechanical Urticaria (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT04428476/Prot_002.pdf
  • Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT04428476/SAP_001.pdf